CLINICAL TRIAL: NCT03742934
Title: Evaluation of Short Peptide Formula for Bowel Preparation in Video Capsule Endoscopy
Brief Title: Short Peptide Formula for Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, The director of gastroenterology of Children's Hospital of Fudan University, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PreparationVCE
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Capsule Endoscopy; Pediatric Disorder
Keywords: Bowel preparation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formula group (Experimental): short peptide formula prior to capsule endoscopy
  Interventions: Other: Short peptide
- Control group (Other): regular liquid diet
  Interventions: Other: Liquid diet

INTERVENTIONS:
Other: Short peptide — Short peptide formula during bowel preparation
  Arms: Formula group
Other: Liquid diet — Liquid diet during bowel preparation
  Arms: Control group

SUMMARY:
Video capsule endoscopy (VCE) is a noninvasive diagnostic tool used to assess the small bowel pathology. The diagnostic value of VCE is mostly dependent on the cleanliness of the colon. Investigators are aimed to prospectively assess the quality of bowel preparation in pediatric patients receiving short peptide diet versus those receiving liquid diet.

ELIGIBILITY:
Inclusion Criteria:

* Indications of capsule endoscopy;
* Informed consent form obtained.

Exclusion Criteria:

* Contraindication of capsule endoscopy;
* Unwilling to participate;
* Formula allergy;
* Unable to swallow the capsule.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Cleansing score | assessed through study completion, an average of 1 year
  Cleansing scores were recorded according to a predetermined criterion

SECONDARY OUTCOMES:
Diagnostic yield | assessed through study completion, an average of 1 year
  Percentage of positive cases
Completion rate | assessed through study completion, an average of 1 year
  CE was considered complete when the cecum was reached within recording time

OTHER OUTCOMES:
Adverse events | assessed through study completion, an average of 1 year
  Adverse events
Bristol scores | assessed through study completion, an average of 1 year
  average Bristol scores during bowel preparation

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, PhD, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goyal J, Goel A, McGwin G, Weber F. Analysis of a grading system to assess the quality of small-bowel preparation for capsule endoscopy: in search of the Holy Grail. Endosc Int Open. 2014 Sep;2(3):E183-6. doi: 10.1055/s-0034-1377521. Epub 2014 Jul 16. PMID 26134966
- [Background] van Tuyl SA, den Ouden H, Stolk MF, Kuipers EJ. Optimal preparation for video capsule endoscopy: a prospective, randomized, single-blind study. Endoscopy. 2007 Dec;39(12):1037-40. doi: 10.1055/s-2007-966988. PMID 18072052